CLINICAL TRIAL: NCT02049489
Title: Immunological Targeting of CD-133 in Recurrent Glioblastoma: A Multi-center Phase I Translational and Clinical Study of an Autologous CD-133 DC Vaccine
Brief Title: A Study of ICT-121 Dendritic Cell Vaccine in Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Precision Life Sciences Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICT-121 DC-01
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Glioblastoma Multiforme
Keywords: ICT-121; glioblastoma; immunotherapy; dendritic cell vaccine; CD133
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICT-121 DC vaccine (Experimental): Autologous dendritic cells pulsed with peptide antigens
  Interventions: Biological: ICT-121 DC vaccine

INTERVENTIONS:
Biological: ICT-121 DC vaccine — autologous dendritic cells pulsed with peptide antigens

SUMMARY:
This study will evaluate a type of immunotherapy in which the patient's immune system will be stimulated to kill tumor cells. ICT-121 dendritic cell (DC)vaccine is made from patient's white blood cells. This vaccine will be tested in patients with recurrent glioblastoma to assess safety, tolerability and clinical response. Patient's white blood cells (WBC) will be collected from blood and cultured to yield autologous DC. The DC will be mixed with purified peptides from the CD133 antigen. The DC vaccine will be given back to the patient over several months. The goal is to stimulate the patient's immune system to CD133 to kill the patient's glioblastoma tumor cells.

DETAILED DESCRIPTION:
Immunotherapy holds promise in oncology for the potential to provide targeted anti-tumor therapy with minimal adverse events. The goal of this study is to assess immunotherapy directed to CD133 in an autologous dendritic cell product called ICT-121. CD133 antigen is overexpressed on many types of cancer cells and is associated with shortened survival. CD133 positive cancer stem cells are resistant to chemotherapy. Patients with recurrent glioblastoma who have the HLA A2 phenotype will receive autologous vaccine of DC pulsed with purified peptides from CD133.

Approximately 20 patients with any recurrence of glioblastoma multiforme (GBM) will be treated. After informed consent and screening, patients will undergo apheresis to collect peripheral blood mononuclear cells (PBMCs). Monocytes will be purified and cultured into dendritic cells (DC) that are pulsed with purified peptides from CD133 antigen. The pulsed dendritic cells will then be aliquoted and frozen. Patients will have the autologous DCs reinfused intradermally. Patients will receive at least four intradermal injections of the autologous DC vaccine and additional vaccines during a maintenance phase. The goal is to induce a cytotoxic T cell response to CD133 positive cells. The primary objective of the study is to assess safety and tolerability. Clinical response rates will be monitored as well as the immune responses to CD133.

ELIGIBILITY:
Inclusion Criteria:

1. Any recurrence of a glioblastoma multiforme
2. ≥ 18 years of age
3. Human leukocyte antigen HLA A2 positive
4. Karnofsky Performance Score (KPS) of ≥ 70%
5. Baseline hematologic studies and chemistry profiles must meet the following criteria:

   * hemoglobin (Hgb) > 9.9 g/dL
   * absolute neutrophil count (ANC) > 1000/mm3
   * platelet count > 100,000/mm3
   * blood urea nitrogen (BUN) < 30 mg/dL
   * creatinine < 2 mg/dL
   * alkaline phosphatase (ALP), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 4x upper limit of normal (ULN)
   * prothrombin time (PT) and activated partial thromboplastin time (PTT) ≤ 1.6 x control unless therapeutically warranted
6. Female patients of child bearing potential must have negative serum pregnancy test
7. If not surgically sterile, male and female patients of childbearing age must use double barrier contraception (hormonal; intrauterine device; barrier)
8. Written informed consent, Release of Medical Records Form and HIPAA reviewed and signed by patient or legally authorized representatives
9. Ability to understand and the willingness to sign a written informed consent document.
10. Any Grade 3 or 4 toxicities (according to NCI CTCAE) resolved for at least 2 weeks prior to first treatment

Exclusion Criteria:

1. Radiosurgery including Gamma Knife, linear accelerator based radiosurgery, CyberKnife and placement of Gliadel wafer
2. Presence of any other active malignancy or prior history of malignancy, except for: basal cell carcinoma of the skin, cervical carcinoma in situ, early stage prostate carcinoma not requiring active treatment
3. New York Heart Association >/= Grade 3 congestive heart failure within 6 months prior to study entry
4. Uncontrolled or significant cardiovascular disease, including:

   * Myocardial infarction and transient ischemic attack or stroke within 6 months prior to enrollment
   * Uncontrolled angina within 6 months
   * Diagnosed or suspected congenital long QT syndrome
   * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes);
   * Clinically significant abnormality on electrocardiogram (ECG)
5. Pulmonary disease including or greater than grade 2 dyspnea or laryngeal edema, grade 3 pulmonary edema or pulmonary hypertension according to CTCAE 4.03
6. Severe acute or chronic medical or psychiatric condition that could increase the risk associated with trial participation or trial drug administration or could interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into the trial. This includes but is not limited to the following:

   1. Immunosuppressive disease
   2. Chronic renal disease / failure
   3. Concurrent neurodegenerative disease,
   4. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of the protocol.
7. Presence of an acute infection requiring active treatment with antibiotics/antivirals; prophylactic administration is allowed
8. Known history of an autoimmune disorder
9. Known human immunodeficiency virus positivity or acquired immunodeficiency syndrome related illness or other serious medical condition
10. Breastfeeding
11. Received any other therapeutic investigational agent within 30 days of screening, except for immunotherapy. Patients with previous immunotherapy are not eligible regardless of timing.
12. Contraindication to MRI
13. Foreseeable condition which would preclude the reduction of steroids (dexamethasone) to a maximum of 2 mg BID within a week prior to apheresis -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of an autologous ICT-121 DC vaccine | 2-3 years
  To assess safety of the autologous ICT-121 DC vaccine the following will be monitored: Serious Adverse events, treatment emergent adverse events, treatment related toxicities

SECONDARY OUTCOMES:
Response rate and immune response to autologous ICT-121 DC vaccine | 2-3 years
  The following parameters for response rate and immune response will be measured:
  The rates of OS and PFS assessed every 2 months until the end of the study; Health-related quality of life parameters in patients treated as above; Post vaccination biopsy/resection (optional) - Assess antigen expression; Overall response rate, defined as the percentage of patients showing either partial response or complete response, will be assessed in patients with measurable disease on MRI; Predictors of response; Immune Response (cytotoxic T-Cell response) to the ICT-121 DC vaccine epitopes.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Gringeri, Ph.D., Study Director — Precision Life Sciences Group
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - JFK New Jersey Neuroscience Institute, Edison, New Jersey
  - Penn State Hershey Neuroscience Institute, Hershey, Pennsylvania
  - Baylor Research Institute - Charles A. Sammons Cancer Center, Dallas, Texas